CLINICAL TRIAL: NCT02733848
Title: A Proof-of-Concept Study Using Pancreatic Enzyme Replacement for the Treatment of Post-Roux-en-Y Gastric Bypass Hypoglycemia
Brief Title: CREON for the Treatment of Post-RYGB Hypoglycemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Moahad S Dar, Clinical Associate Professor of Medicine, Division of Endocrinology & Metabolism, East Carolina University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UMCIRB 11-001311
Record Dates: First submitted 2016-02-15; First posted 2016-04-12 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Hypoglycemia
Keywords: Roux-en-Y gastric bypass; Hypoglycemia; Creon
MeSH Terms: conditions — Hypoglycemia | interventions — Pancrelipase; Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- DIET (Experimental): A registered dietician (RD) will meet with and thoroughly review the patients diet. The patient will be counseled on a diet lower in refined carbohydrates and higher in protein.
  Interventions: Other: Diet
- Creon (Active Comparator): Subjects will be provided Creon at a dose of 500 units/kg of lipase to be taken with meals and snacks to see if this decreases frequency and severity of hypoglycemia.
  Interventions: Drug: Creon
- Placebo (Placebo Comparator): Subjects will be provided placebo and advised to take it with meals and snacks to provide.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Creon — Creon is a porcine derived pancreatic enzyme supplement that comes in in fixed dose combinations of lipase, protease, and amylase, respectively. Dosing is based on lipase per kilograms per meal (i.e. lipase units/kg/meal). Subjects will be started at a dose of 500 units of lipase/kg/meal and snacks at week 4 and continued until week 8. A follow-up visit at week 6 will assess patient for tolerance to Creon and need for dosage adjustment.
  Formulations come in different fixed dose combinations as follows:
  Creon: Lipase 3000 USP units, protease 9500 USP units, and amylase 15,000 USP units
  Creon: Lipase 6000 USP units, protease 19,000 USP units, and amylase 30,000 USP units
  Creon: Lipase 12,000 USP units, protease 38,000 USP units, and amylase 60,000 USP units
  Creon: Lipase 24,000 USP units, protease 76,000 USP units, and amylase 120,000 USP units
  Creon: Lipase 36,000 USP units, protease 114,000 USP units, and amylase 180,000 USP units
  Arms: Creon
Other: Diet — A registered dietician will meet with the subject and take a thorough review of the patient's dietary history. The subject will then be counseled on a lower carbohydrate and higher protein diet. This diet will be continued for the entire 12 week of the study. The registered dietician will reinforce dietary recommendations by phone on week 2, 4 and 8, respectively.
  Arms: DIET
Other: Placebo — Placebo will be given to the patient in single blind fashion with the subject unaware but PI aware of study drug assignment from week 8-12. Placebo tablets will be given with meals and snacks similar to CREON to maintain patient blinding to study drug assignment. A follow-up visit on week 10 to review patient tolerance, side effects and possible drug adjustment.
  Arms: Placebo

SUMMARY:
Hypoglycemia is an increasingly recognized complication of Roux-en-Y gastric bypass (RYGB) that is poorly understood and difficult to treat. Investigators hypothesize that after RYGB some patients have incomplete carbohydrate absorption in the small intestine which leads to inconsistent glucose levels and hypoglycemia during oral consumption of a meal. Investigators further hypothesize that pancreatic enzyme supplementation with (Creon) during meals and snacks will improve carbohydrate absorption and lead to more stable glucose levels in patients with post-RYGB hypoglycemia.

DETAILED DESCRIPTION:
Primary Objective: Evaluate the feasibility and safety of Creon in the treatment of post-RYGB hypoglycemia as add-on therapy to a diet higher in protein and lower in carbohydrate.

Secondary Objective: Evaluate utility of continuous glucose monitoring (CGM) in monitoring hypoglycemia as an adjunct to standard venous blood testing using a glucometer in post-RYGB hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years and older
* At least 6 months post-RYGB surgery
* Clinical history of post-surgical hypoglycemia evident by subjective symptoms (i.e. tachycardia, sweating, hunger, confusion) and glucose monitoring demonstrating a venous blood sugars < 70 mg/dL
* Women must be postmenopausal, surgically sterile, not heterosexually active or heterosexually active using highly effective method of birth control
* Women of childbearing potential must have negative pregnancy test
* Subjects must have signed an informed consent document indicating they understand the purpose of and procedures required for the study and be willing to participate in the study
* Willing and able to adhere to restrictions and follow instructions specific to this study
* Adequate compliance in performing self-monitoring blood glucose (SMBG) testing at least three or more times per week and taking assigned medication dose as instructed

Exclusion Criteria:

* Current or past history of type 1 or type 2 diabetes
* Known hypersensitivity to Creon
* Known hypersensitivity to pork-derived products
* Liver function studies 2 times the upper limit of normal (ALT & AST) and/or a GFR < 90
* History of fibrosing colonic strictures
* History of gastroparesis, dysphagia, chronic abdominal pain, gastric outlet obstruction, chronic pancreatitis
* History of stomach, small intestine or colon surgery other than Roux-en-Y gastric bypass
* An active cancer of any type requiring concurrent treatment
* History of gout or hyperuricemia
* Current anemia requiring iron replacement
* Any clinically significant condition that in the opinion of the investigator would make participation not in the best interest or safety of the subject or could prevent limit or confound the specific endpoints assessments
* Not participating in any other research study
* Known history of drug or alcohol abuse within 6 months of screening visit
* Pregnancy or lactation (breastfeeding)
* Informed consent withdrawal by subject

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Frequency of Hypoglycemia | 2 years
  The effect of DIET, CREON and PLACEBO on the number of hypoglycemic events (i.e. <70 mg/dl) will be assessed using a standard blood glucose monitor that measures glucose in venous blood.

SECONDARY OUTCOMES:
Continuous Glucose Monitoring using the Medtronic iPro 2 | 2 years
  The effect of DIET, CREON and PLACEBO on the percent of time iPro 2 glucose values are less than 70 mg/dL will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Moahad S Dar, MD, Principal Investigator — Brody School of Medicine at East Carolina University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sarwar H, Chapman WH 3rd, Pender JR, Ivanescu A, Drake AJ 3rd, Pories WJ, Dar MS. Hypoglycemia after Roux-en-Y gastric bypass: the BOLD experience. Obes Surg. 2014 Jul;24(7):1120-4. doi: 10.1007/s11695-014-1260-8. No abstract available. PMID 24737312